CLINICAL TRIAL: NCT05522439
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Phase II Clinical Study to Evaluate the Pharmacodynamic, Efficacy and Safety of Multiple Subcutaneous Injections of SHR-1703 in Asthma Patients With Eosinophil Phenotype
Brief Title: A Study to Evaluate the Pharmacodynamic, Efficacy and Safety of SHR-1703 in Asthma Patients With Eosinophil Phenotype
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1703-201
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Asthma With Eosinophilic Phenotype

STUDY DESIGN:
Intervention Model Description: Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Phase II Clinical Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Subjects receiving SHR-1703 dose 1 (Experimental)
  Interventions: Drug: SHR-1703; Drug: SHR-1703 Placebo
- Subjects receiving SHR-1703 dose 2 (Experimental)
  Interventions: Drug: SHR-1703
- Subjects receiving SHR-1703 dose 3 (Experimental)
  Interventions: Drug: SHR-1703; Drug: SHR-1703 Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: SHR-1703 Placebo

INTERVENTIONS:
Drug: SHR-1703 — SHR-1703 will be administered by SC injection.
  Arms: Subjects receiving SHR-1703 dose 1; Subjects receiving SHR-1703 dose 2; Subjects receiving SHR-1703 dose 3
Drug: SHR-1703 Placebo — Matching Placebo will be administered by the SC route.
  Arms: Placebo; Subjects receiving SHR-1703 dose 1; Subjects receiving SHR-1703 dose 3

SUMMARY:
The purpose of this study is to evaluate the Pharmacodynamic, Efficacy and Safety of SHR-1703 in Asthma Patients with Eosinophil Phenotype.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75years (inclusive).
2. Weight ≥40 kg.
3. History of asthma≥ 1 year.
4. Documented treatment with Medium or high daily dose inhaled corticosteroid with additional controller medication within the 3 months prior to randomization.
5. Previously confirmed history of one or more asthma exacerbations within 1 year prior to randomization.
6. Blood eosinophils of ≥150 cells/µL at screening and baseline.
7. Pre-Bronchodilator FEV1% pred≥40% and<80% at screening and baseline.
8. Asthma Control Questionnaire-6 score≥1.5.
9. Use highly effective contraceptive measures.
10. Willing to sign the informed consent form to participate in this study.

Exclusion Criteria:

1. Subjects with Clinically significant pulmonary diseases；
2. Subjects with other diseases that could lead to elevated eosinophils；
3. Subjects with Immunodeficiency；
4. Poorly controlled hypertension;
5. Subjects with severe cerebrovascular disease;
6. Subjects with infection history requiring clinical intervention；
7. Subjects with parasitic infection；
8. Diagnosed Malignant tumor within 5 years prior to randomization;
9. Used non-selective β-blockers within 1 week prior to randomization;
10. Used either 5-lipoxygenase inhibitor or Phosphodiesterase-4 inhibitor within 1 week prior to randomization;
11. Blood donation or massive blood loss, or transfusion of blood products or immunoglobulins within 4 weeks prior to randomization;
12. Live attenuated vaccine inoculated within 4 weeks before randomization;
13. Allergen Immunotherapy within 8 weeks prior to randomization；
14. Used systemic immunosuppressants or immunomodulators, or biologics or Th2 cytokine inhibitors within 12 weeks prior to randomization or within 5 half-lives of the drug;
15. Bronchial thermoplasty within 1 year prior to randomization；
16. Subjects have planned Surgery or other medical procedures that may affect evaluation during the study period;
17. Subjects with significant laboratory abnormality at screening；
18. Subjects have prolonged QTc interval or other electrocardiogram abnormality with significant safety risk at screening;
19. Current smokers or ex-smokers who have given up smoking for <6 months ，or positive smoke test, and/or have a smoking pack history of > 10 pack years;
20. History of drug or substance abuse or alcohol abuse within 1 year prior to screening;
21. Subjects participated another clinical studies and received active drug within 30 days or 5 half-lives prior to screening;
22. Subjects is pregnant, lactating,or planning to become pregnant;
23. Subjects have a known history of hypersensitivity or intolerance to anti-IL-5 mabs or other biological agents;
24. Other conditions unsuitable for participation in the study per investigator judgement.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in Blood Eosinophils | Up to Week 52

SECONDARY OUTCOMES:
Changes from baseline in Pre- and post-Bronchodilator FEV1 | Up to Week 52
Changes from baseline in Pre- and post-Bronchodilator FEV 1% pred | Up to Week 52
Changes from baseline in Pre- and post-Bronchodilator FVC | Up to Week 52
Changes from baseline in Pre- and post-Bronchodilator PEF | Up to Week 52
Changes from baseline in n fractional exhaled nitric oxide (FeNO) | Up to Week 52
Changes from baseline in Asthma Control Questionnaire-6(ACQ-6) | Up to Week 52
Changes from baseline in Standardized Asthma Quality of Life Questionnaire (AQLQ) | Up to Week 52
Frequency of use of asthma relievers | Up to Week 24
Frequency of exacerbations of asthma | Up to Week 24
Frequency of severe exacerbations of asthma | Up to Week 24
Time to first exacerbation of asthma | Up to Week 24
Time to first severe exacerbation of asthma | Up to Week 24

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided